CLINICAL TRIAL: NCT05585437
Title: Effect of Gastric Cancer Specialist Training Program in Laparoscopic Gastric Cancer Surgery: a Survey Based on Follow-up Questionnaire
Brief Title: Effect of Gastric Cancer Specialist Training Program in Laparoscopic Gastric Cancer Surgery（STP-LRG-1）
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Clinical Professor, Fujian Medical University
Other Study IDs: FUGES-026
Record Dates: First submitted 2022-02-22; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- gastric cancer specialist training program
  Interventions: Procedure: gastric cancer specialist training program

INTERVENTIONS:
Procedure: gastric cancer specialist training program — The gastric cancer specialist training program includes technical training and non-technical training. The technical training includes 1. The whole process of laparoscopic gastric cancer surgery technical teaching 2. Operation practice 3. Operation video review, non-technical training includes 1. Difficult case discussion 2. Specialists Session 3. Lymph node sorting training.

SUMMARY:
To prospectively evaluate the effect of the gastric cancer specialist training program of Fujian Medical University Union Hospital on laparoscopic gastric cancer surgery.

DETAILED DESCRIPTION:
Laparoscopic gastric cancer surgery has the advantages of less trauma, quick postoperative recovery, less postoperative pain symptoms, less postoperative complications, and shorter average hospital stay. In addition, the surgical safety and oncological efficacy of laparoscopic radical gastrectomy for gastric cancer have been obtained. Confirmed by numerous clinical studies.

However, due to the difficult operation, complex anatomy and high technical requirements of laparoscopic gastric cancer surgery, the operator needs to have rich experience in laparotomy, skilled laparoscopic operation skills, and the ability to actively prevent and deal with complications after surgery. Therefore, at this stage, laparoscopic radical gastrectomy for gastric cancer is only suitable for large hospitals with certain conditions, and it should be gradually carried out on the basis of chief surgeons with rich clinical experience in radical gastrectomy and skilled laparoscopic technical experience.

The gastric cancer specialist training program (STP-LRG-1) of Fujian Medical University Affiliated Union Hospital (STP-LRG-1) has more than 9 years of trainee training experience. The effectiveness of STP-LRG-1 has not been prospectively evaluated, so this study aimed to prospectively evaluate whether STP-LRG-1 can improve the surgical skills of trainees and ultimately improve short-term outcomes for patients during and after surgery

ELIGIBILITY:
Inclusion Criteria:

1. The title of fellow physician or above, with experience in performing laparoscopic radical gastrectomy for gastric cancer independently or under supervision;
2. The hardware facilities and staffing of the operating room support the completion of laparoscopic gastric cancer surgery;
3. Surgical videos of laparoscopic radical gastrectomy before and after the training required for this study can be provided;
4. Clinicopathological data, intraoperative and postoperative short-term outcome data of the patients operated by the surgeon before and after training can be provided;
5. Informed consent

Exclusion Criteria:

1. Refuse to carry out laparoscopic gastric cancer surgery;
2. Due to the limitations of equipment or policies, the unit cannot routinely carry out laparoscopic gastric cancer surgery;
3. Those who have not performed laparoscopic gastric cancer surgery within 1 month before participating in the training and cannot provide video;
4. Those who are not expected to perform laparoscopic gastric cancer surgery within 1 month after participating in the training;
5. Participate in other clinical investigators during the same period.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants were gastric cancer specialists who trained in the Department of Gastric Surgery of FJMU-UH from 2013 to 2020
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
patient complication rate | one year
  Rate of reduction in surgical patient complications after trainee training

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China